CLINICAL TRIAL: NCT03888768
Title: ProPBM : A Randomised Control Trial Comparing a Modified Patient Blood Management Protocol Against Standard Care for Patients Undergoing Major Surgery
Brief Title: ProPBM : A Modified Patient Blood Management Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Tan Jenq Uei, Trainee of Master of Anaesthesiology University of Malaya, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46050
Record Dates: First submitted 2019-03-01; First posted 2019-03-25 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Iron-deficiency
Keywords: intravenous iron isomaltoside(monofer); iron deficiency; anaemia; patient blood management
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Anemia

STUDY DESIGN:
Intervention Model Description: ProPBM arm and standard Care arm
Masking Description: patient will be randomised into ProPBM and standard care arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProPBM (Active Comparator): Pre-operative: patient will be screened for iron deficiency and anemia and administered IV monofer Intra-operative:IV tranexamic Acid 1gm will be administered at the beginning of surgery and blood transfusion triggered by Allowable blood loss Post-operative: IV Iron monofer will be given to those with estimated blood loss >1L and subsequent post operative follow up till 6month
  Interventions: Drug: MonoFer
- Standard Care (No Intervention): patient will received standard hospital practise

INTERVENTIONS:
Drug: MonoFer — Administration of IV Monofer will be given according to body weight as recommended by the drug manufacturer.
  Other Names: isomaltoside
  Arms: ProPBM

SUMMARY:
The introduction of a modified perioperative patient blood management protocol with intravenous iron intervention for iron deficiency anaemic patients would reduce the need for allogenic blood transfusion and reduce perioperative morbidity and mortality.

DETAILED DESCRIPTION:
Patient blood management (PBM), refers to "the timely application of evidence based medical and surgical concepts designed to maintain haemoglobin concentration, optimise haemostasis and minimize blood loss in an effort to improve patient outcome.

PBM relies on three corresponding aspects:

1. Optimising haemopoiesis,
2. Minimising bleeding and blood loss
3. Harnessing and optimising physiological tolerance of anaemia.

Therefore, this randomised control trial aims to study the effect of applying a modified patient blood management protocol on the perioperative allogenic blood transfusion incidence, mortality and morbidity in patients undergoing major surgery in gynaecology, intraabdominal surgery and orthopaedics comparing with current practice.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing major surgery in gynaecology, gastrointestinal surgery and orthopaedics
* Major surgery defined as either Intrabdominal surgery or main joint surgery, Risk of blood loss >15% blood volume
* Aged between 18 to 80 years of age
* The patient must be willing and able to provide written informed consent for the study

Exclusion Criteria:

* Allergy or known sensitivity to parenteral iron
* Hypersensitivity to the active substance, Iron(III) Isomaltoside or any of its excipients listed in the summary of product characteristics
* Patients with iron overload

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative allogenic blood transfusion. | Participants will be followed from date of hospital entry until date of discharge up to 6 months
  To assess the incidence of allogenic blood transfusion occurring within the total length of hospital stay within the same admission of a surgical procedure performed under general or regional anaesthesia

SECONDARY OUTCOMES:
Change in haemoglobin (Hb) concentrations from baseline | Preoperative basline and one day before surgery after MonoFer administration expected up to 2 weeks
  To assess the extent of increase in preoperative hemoglobin levels(baseline) and hemoglobin level one day before surgery, after the administration of IV MonoFer in ProPBM arm
Quality of Life of patient | preoperative (baseline), one month, six month
  To assess patient's quality of life using Short Form (12) Health Survey(SF-12) is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight domain scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Postoperative Morbidity | Day one postoperative, postoperative one week,postoperative one month, postoperative six month
  To assess postoperative morbidity using Postoperative Morbidity Survey(POMS).Patients are assessed for diagnostic features in nine domains (pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, haematological, wound and pain). For each domain, either presence or absence of morbidity is recorded on the basis of objective criteria.
Mortality rate | Participants will be followed up expected till 6 months
  To assess the incidence of mortality after surgery in both ProPBM arm and standard arm
Total hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Participants will be followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ng, Principal Investigator — UMMC
Locations (1):
- University Malaya Medical Centre, Jalan Universiti, Kuala Lumpur, Kuala Lumpur, Malaysia